CLINICAL TRIAL: NCT04275908
Title: Classification and Assessment of Mental Health Performance Using Schematics
Acronym: CAMPUS
Status: Completed | Type: Observational
Sponsor: Clarigent Health (Industry)
Collaborators: Children's Hospital Medical Center, Cincinnati (Other); University of Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 102-2019
Record Dates: First submitted 2020-01-31; First posted 2020-02-19 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Suicide Ideation; Suicidal Intention; Suicide and Depression
MeSH Terms: conditions — Suicide; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: MHSAFE app — App to detect presence of mental state

SUMMARY:
This is an open enrollment study to collect data for the optimization of smartphone-based algorithms for the early detection of mental health and suicidal risk in a student population. Approximately 2000 students, ages 8-23, will be recruited by therapists across 30 schools and mental health centers.

ELIGIBILITY:
Inclusion Criteria:

* Currently a client receiving services from mental health agency at a school or outpatient, or at a college/university counseling center
* Age ≥ 8 years and < 23years
* Able to provide informed consent, parental permission or assent
* English as a primary language

Exclusion Criteria:

* Participants with communication disorders (linguistic or articulation)
* Any minor participants for whom parental or legal guardian consent cannot be obtained.
* History of any other serious medical or psychiatric condition that would interfere with the ability of the patient to complete the study or would make it ethically unfeasible to enroll them
* Participants with an intellectual disability that the therapist deems a barrier to participation

Ages: 8 Years to 23 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Thirty sites across Southwest Ohio will be recruited, including schools (using the school-based therapists), community mental health centers, and colleges/universities (counseling centers). Approximately 150 therapists across 30 sites will be recruited to enroll students from their current caseloads.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-01-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Algorithm development | 3 years
  Participants will be asked about their mental health using standardized questionnaires and a specific set of additional questions developed to encourage an open conversation with the therapist. The app will record the therapy session and a proprietary algorithm will be tested to determine if it can accurately detect the presence of a mental state (for example, suicidal intention) as compared with the standardized questionnaires (e.g. Columbia scale) and the therapists' clinical impression.
App optimization | 3 years
  Convenient and accessible use of the app in a variety of settings where adolescents and young adults may require intervention for mental health and suicide-related concerns. Upon completion of the therapy sessions, the therapists will be asked to complete a questionnaire to provide feedback on the usability of the device in a real-world setting. This information will drive modifications to the app and to the device that it is used with (e.g. smartphone, tablet) to create second generation models that are user-friendly and provide valuable information in clinical settings.

CONTACTS AND LOCATIONS:
Overall Officials: Lesley Rohlfs, Study Director — Clarigent Health
Locations (1):
- Clarigent Health, Mason, Ohio, United States

IPD SHARING:
Plan to Share IPD: No